CLINICAL TRIAL: NCT03102658
Title: Micafungin (Mycamine®) Pharmacokinetics Given as a Single Intravenous Dose to Obese Patients (MICADO).
Brief Title: Micafungin Pharmacokinetics in Obese Patients
Acronym: MICADO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: St. Antonius Hospital (Other); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UMCN-AKF 16.02
Record Dates: First submitted 2017-01-05; First posted 2017-04-06 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2017-09

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Obese subjects 100mg (Experimental): 8 subjects with a BMI>40kg/m2 will receive 100mg Micafungin
  Interventions: Drug: Micafungin
- Obese subjects 200mg (Active Comparator): 8 subjects with a BMI>40kg/m2 will receive 200mg Micafungin
  Interventions: Drug: Micafungin
- non-obese subjects (Active Comparator): 8 non obese subjects with a BMI >18.5 and <25 kg/m2 will receive 100mg Micafungin
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — Administration of study drug
  Other Names: Mycamine

SUMMARY:
Because micafungin is generally well tolerated and appears to have limited interaction with other drugs, it is a potential important agent in the treatment of invasive fungal infections. Although micafungin is approved for the treatment of invasive candidiasis, dosing guidelines for micafungin in (morbidly) obese patients are not available. Subsequently, the pharmacokinetic profile of micafungin (as well as other echinocandins) in this specific patient population is still largely unknown.

To build a valid pharmacokinetic model, obese patients with a BMI ≥ 40 undergoing endoscopic gastric bypass surgery will receive a single dose of 100 mg or 200mg micafungin (besides standard anti-bacterial prophylaxis) and samples for a pharmacokinetic curve will be taken. These PK-values can then be compared to the PK in a normal-weight group which will receive 100mg micafungin

DETAILED DESCRIPTION:
Obese patients with a BMI ≥ 40 kg/m2 undergoing endoscopic gastric bypass surgery will receive a 100 mg or a 200mg dose of micafungin. A PK curve will be determined after administration at t=0.5, 0.95, 1.25, 1.5, 2, 4, 8, 12, 24, and (if feasible) 48 hours post infusion. Blood samples (4 mL) on PK days will be taken to obtain at least 2.0 mL of plasma.

ELIGIBILITY:
Inclusion Criteria

1. Subjects BMI:

   * obese groups: subject must have a BMI > 40 kg/m2 at the time of inclusion,
   * non-obese group: subject must have a BMI ≥18.5 and < 25kg/m2 at the time of inclusion.
2. Subject is at least 18 of age on the day of screening and not older than 65 years of age on the day of dosing;
3. If a woman, is neither pregnant nor able to become pregnant and is not nursing an infant;
4. Subject is able and willing to sign the Informed Consent before screening evaluations.

   For the non-obese subjects the following additional exclusion criteria apply:
5. Subject is in good age-appropriate health condition as established by medical history, physical examination, electrocardiography, results of biochemistry, hematology and urinalysis testing within 4 weeks prior to study drug administration. Results of biochemistry, hematology and urinalysis testing should be within the laboratory's reference ranges. If laboratory results are not within the reference ranges, the subject is included based on the investigator's judgment that the observed deviations are not clinically relevant. This should be clearly recorded;
6. Subject has a normal blood pressure and pulse rate, determined by the investigator;
7. Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to study drug administration.

Exclusion Criteria:

1. Documented history of sensitivity to medicinal products or excipients similar to those found in the micafungin preparation;
2. History of, or known abuse of drugs, alcohol or solvents (up until a maximum of three months before study drug administration);
3. Inability to understand the nature of the trial and the procedures required;
4. Use of medication that has known interaction with study drug as determined by the investigator up to 4 weeks prior to study drug administration.

   For the non-obese subjects the following additional exclusion criteria apply:
5. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs or clinical laboratory determinations;
6. Clinical relevant liver enzymes (alkaline phosphatase, alanine aminotransferase, aspartate transaminase) abnormalities at screening;
7. Donation of blood or plasma to a blood bank or in a clinical study (except a screening visit) within 4 weeks prior to study drug administration;
8. Blood transfusion within 8 weeks prior to study drug administration;
9. Inability to be venipunctured and/or tolerate venous access;
10. Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), psychiatric disorders, gastro-intestinal disorders, renal disorders, hepatic disorders (Child-Pugh B or C), hormonal disorders (especially diabetes mellitus), coagulation disorders;
11. Any other sound medical, psychiatric and/or social reason as determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Micafungin concentration in plasma to examen the area under the plasma concentration versus time curve (AUC0-48) | Up to 3 months
  The exposure to micafungin in obese will be compared with that in non-obese subjects.

SECONDARY OUTCOMES:
Long-term exposure to micafungin after repeated dose | Up to 6 months
  Predict long-term exposure (AUC0-tau) after repeated dosing by popPK modeling and simulation.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Brüggemann, PharmD, PhD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - St Antoniusziekenhuis, Nieuwegein
  - Radboudumc CRCN, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wasmann RE, Smit C, Ter Heine R, Koele SE, van Dongen EPH, Wiezer RMJ, Burger DM, Knibbe CAJ, Bruggemann RJM. Pharmacokinetics and probability of target attainment for micafungin in normal-weight and morbidly obese adults. J Antimicrob Chemother. 2019 Apr 1;74(4):978-985. doi: 10.1093/jac/dky554. PMID 30649375
- See also: paper — https://pubmed.ncbi.nlm.nih.gov/30649375/